CLINICAL TRIAL: NCT02170857
Title: A Randomized Controlled Trial to Evaluate the Effect of Hyaluronic Acid on Infra-bony Defects: A Radiographic and Clinical Study.
Brief Title: Effect of Hyaluronic Acid in the Treatment of Periodontal Pockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Perio-05-2014
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Chronic Periodontitis With Infra-bony Defects
Keywords: Hyaluronic acid; infra-bony defects; chronic periodontitis; experimental; radiographic; clinical; periodontal surgical treatment; open flap curettage
MeSH Terms: conditions — Chronic Periodontitis | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open Curettage Only (No Intervention): patients will be treated by the conventional surgical method, i.e. open curettage without injecting any material.
- Open Curettage with Hyaluronic Acid (Experimental): Hyaluronic Acid injection will be employed in conjunction with the ordinary surgical procedure.
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Drug: Hyaluronic Acid — This material will be used in conjunction with the ordinary surgical procedure
  Arms: Open Curettage with Hyaluronic Acid

SUMMARY:
The aim of this study is to evaluate the effect of hyaluronic acid in the surgical treatment of periodontal pockets in people with gum disease.

This research consists of clinical and radiographic studies. Participants should have symmetric periodontal pockets in the upper or lower jaw.

Participants will be treated surgically using hyaluronic acid on one side of the jaw.

Clinical indexes and radiographic cone-beam computed tomographic (CBCT) images will be taken for each participant before surgical treatment and 12 months after surgical treatment.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of hyaluronic acid in the surgical treatment of infra-bony pockets in chronic periodontitis patients.

This research consists of clinical and radiographic studies.

1- The clinical study: is a randomized controlled trial with a split mouth technique.

Chronic periodontitis patients with Infra-bony pockets will be collected from the Department of Periodontics in faculty of dentistry - Damascus university.

Participants should have symmetric infra-bony pockets in the upper or lower premolar area with pocket probing depth more than 6 mm.

Participants will be treated surgically using open flap curettage.

Open flap curettage will be done for each patient in both sides of the jaw, but hyaluronic acid will be used in one of the two sides with random allocation of the site that in going to be treated with hyaluronic acid.

Plaque index, gingival index, bleeding on probing, tooth mobility index, pocket probing depth and clinical attachment loss will be taken for each participant four times; before surgical treatment, 3 months, six months and 12 months after surgical treatment.

Radiographic study: will be done using CBCT radiography technique. CBCT will be taken for each participant before and after 12 months of surgical treatment. Different distances, vertical bone fill and depth of infra-bony defect will be measured on CBCT images.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic periodontitis
* Symmetric Infra-bony defects with periodontal pocket depth more than 6 mm.
* in upper or lower premolar area.
* All participants will be collected from patients attending department of Periodontology - faculty of dentistry for periodontal disease treatment.
* Males and females.
* 35-65 years old.
* Systematically healthy.
* Accepting to participate in the study. Informed written consent will be required.

Exclusion Criteria:

* A history of previous scaling and root planning in the last 6 months
* Smokers
* Pregnant women
* Diabetes mellitus

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in the Clinical Attachment Loss (CAL) | CAL will be measured at four times in this study: one week before surgical treatment, 3 months post-surgery, six months post-surgery and 12 months post-surgery
  Clinical Attachment Loss (CAL): it is the distance between the cement-enamel junction of the tooth and the bottom of the pocket.
  CAL will be performed using a dental probe.
Vertical bone fill | at 12 months post-surgery
  Vertical bone fill: it is the distance between the base of the infra-bony defect and cement-enamel junction before surgery minus the distance between base of the infra-bony defect and cement enamel junction after surgery.
  It will be measured on CBCT images.

SECONDARY OUTCOMES:
Change in the Pocket Probing Depth (PPD) | PPD will be measured at four times in this study: one week before surgical treatment, 3 months post-surgery, six months post-surgery and 12 months post-surgery
  Pocket Probing Depth (PPD): it is the distance from the gingival margin to the bottom of the pocket at four sites per tooth. PPD will be measured using a dental probe.
Buccolingual distance | at 12 months post-surgery
  Buccolingual distance: is the distance between buccal wall and lingual wall of the infra-bony pocket.
Mesiodistal distance | at 12 months post-surgery
  Mesiodistal distance: is the distance between mesial wall and distal wall of the infra-bony pocket.
Depth of infra-bony defect | at 12 months post-surgery
  Depth of infra-bony defect: is the distance between the base of the infra-bony defect and the most coronal level of alveolar crest.

CONTACTS AND LOCATIONS:
Overall Officials: Lina Bashour, DDS MSc, Principal Investigator — PhD student, Department of Periodontics, University of Damascus Dental School, Damascus; Razan Khattab, DDS MSc PhD, Study Director — Professor of Periodontics, Dean of the Dental School, University of Damascus Dental School, Damascus
Locations (1):
- Department of Periodontics, University of Damascus Dental School, Damascus, Syria

REFERENCES:
- [Background] Baldini A, Zaffe D, Nicolini G. Bone-defects healing by high-molecular hyaluronic acid: preliminary results. Ann Stomatol (Roma). 2010 Jan;1(1):2-7. Epub 2010 Jun 29. PMID 22238698
- [Background] Ballini A, Cantore S, Capodiferro S, Grassi FR. Esterified hyaluronic acid and autologous bone in the surgical correction of the infra-bone defects. Int J Med Sci. 2009;6(2):65-71. doi: 10.7150/ijms.6.65. Epub 2009 Feb 26. PMID 19277251
- [Background] Bansal J, Kedige SD, Anand S. Hyaluronic acid: a promising mediator for periodontal regeneration. Indian J Dent Res. 2010 Oct-Dec;21(4):575-8. doi: 10.4103/0970-9290.74232. PMID 21187628
- [Background] Briguglio F, Briguglio E, Briguglio R, Cafiero C, Isola G. Treatment of infrabony periodontal defects using a resorbable biopolymer of hyaluronic acid: a randomized clinical trial. Quintessence Int. 2013 Mar;44(3):231-40. doi: 10.3290/j.qi.a29054. PMID 23444204
- [Background] Vanden Bogaerde L. Treatment of infrabony periodontal defects with esterified hyaluronic acid: clinical report of 19 consecutive lesions. Int J Periodontics Restorative Dent. 2009 Jun;29(3):315-23. PMID 19537471
- [Background] Gontiya G, Galgali SR. Effect of hyaluronan on periodontitis: A clinical and histological study. J Indian Soc Periodontol. 2012 Apr;16(2):184-92. doi: 10.4103/0972-124X.99260. PMID 23055583